CLINICAL TRIAL: NCT03843502
Title: A Phased Clinical Trial of Dietary Supplemental Kava: Kava Pharmacokinetics
Acronym: KavaPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Thorne HealthTech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201900074 -N; OCR20231 (Other: OnCore); 1R61AT009988-01A1 (NIH); 3R61AT009988-02S1 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Pharmacokinetics
Keywords: kava; dietary supplement; anxiety; generalized anxiety disorder (GAD)
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kava Pharmacokinetics Group (Experimental): Each subject will take three 75 mg kava dietary supplement capsules in a single dose/timepoint and nine blood draws will be collected over an eight hour period following adminstration of kava.
  Interventions: Drug: Kava Dietary Supplement

INTERVENTIONS:
Drug: Kava Dietary Supplement — Participants will be given three 75mg kava capsules.
  Other Names: Kava metabolites

SUMMARY:
Kava is a dietary supplement on the US market and is experiencing a resurgence of its use. Its pharmacokinetic information, however, is lacking which is important for its future effective usage as a dietary supplement or potentially as a botanical therapeutics. This phased trial, based on the recommendation from NIH, is to collect pharmacokinetic data of kava in healthy subjects.

DETAILED DESCRIPTION:
Kava is used in the South Pacific Islands for relaxation and socialization. It is available in the US as a dietary supplement, and was used in Europe in the 1990s to treat mild to moderate anxiety. Some clinical trials suggested kava's efficacy in treating generalized anxiety disorder (GAD), although a recent meta-analysis was inconclusive. While the mechanisms behind kava's anxiolytic activity are not well-established, its clinical use shows no signs of addiction or withdrawal. Kava thus is a promising and potentially novel anxiolytic with a unique mechanism of action. Although kava has been extensively consumed by humans for centuries, its pharmacokinetics have never been characterized in humans. Such knowledge is essential for its future studies of its anxiolytic potential and dose optimization. This study will characterize kava pharmacokinetics, which will set a solid foundation for its future clinical development. To establish kava pharmacokinetics, each participant will take three 75 mg kava capsules in a single dose and the absorption, distribution, metabolism and excretion of kava will be assessed, corresponding to the pharmacokinetic curve. Serum liver biochemistries will then be monitored for up to three months to test liver function response to kava.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Females of potential childbearing status must use adequate contraceptive precautions

Exclusion Criteria:

* Currently taking any medication or supplement other than vitamins
* Inability to refrain from acetaminophen, alcohol, or other potentially hepatotoxic substances during the study
* Have a history of liver disease or currently have liver disease.
* Elevation in serum ALT, AST, ALP or total bilirubin that reaches clinical significance (as determined by the PI) at screening.
* Have an unstable medical, psychiatric, or neurological condition determined by history taken during the screening visit and a physical examination at the baseline visit.
* Have a positive urine drug screen for substances of abuse.
* Currently using tobacco or nicotine containing products of any form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Mathews, MD, Principal Investigator — University of Florida
Locations (1):
- UF CTSI Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruitment for this study via flyers placed in various location in and around the Gainesville area.
Pre-assignment Details: Any individuals who were found to have a positive urine drug screen, had abnormal lab values, or were found to have active suicidal ideation were excluded from the study prior to baseline.
Groups:
- Kava Pharmacokinetics Single Dose Group: 5 subjects will take three 75 mg kava dietary supplement capsules in a single dose/timepoint and nine blood draws will be collected over a twelve hour period following administration of kava.
  Kava Dietary Supplement: Participants will be given three 75mg kava capsules for a total dose of 225mgs.
- Kava Pharmacokinetics 3x a Day Dose Group: 5 subjects will take three 75 mg kava dietary supplement capsules split among three time points during the study visit. Nine blood draws will be collected over a twelve hour study period.
  Kava Dietary Supplement: Participants will be given three 75mg kava capsules for a total dose of 225mgs
Period: Overall Study
Arm/Group | Kava Pharmacokinetics Single Dose Group | Kava Pharmacokinetics 3x a Day Dose Group
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kava Pharmacokinetics Single Dose Group | Kava Pharmacokinetics 3x a Day Dose Group | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 21 [19 to 22] | 21 [18 to 40] | 21 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximum Concentration of Kava in the Blood
Description: Number of hours that it takes for kava metabolites to reach the maximum concentration in the blood based on multiple blood draws over a 12 hour period
Time Frame: pre-dose to 12 hours post-dose
Population: 10 healthy participants were included in the analysis
Measure: Mean (Standard Error); unit: hours
Arm/Group | Kava Pharmacokinetics Single Dose Group | Kava Pharmacokinetics 3x a Day Dose Group
Number analyzed (Participants) | 5 | 5
hours
  Kavain | 1.9 (1.1) | 1.2 (0.8)
  Dihydrokavain | 1.3 (0.9) | 1.2 (0.8)
  Methysticin | 1.9 (1.1) | 1.2 (0.8)
  Dihydromethysticin | 1.5 (1.0) | 1.20 (0.8)
  Yangonin | 1.9 (0.9) | 1.8 (0.8)

ADVERSE EVENTS:
Time Frame: 11 months
Description: Reporting information follows clinicaltrials.gov guidelines
Arm/Group | Kava Pharmacokinetics Single Dose Group | Kava Pharmacokinetics 3x a Day Dose Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kava Pharmacokinetics Single Dose Group (N=5) | Kava Pharmacokinetics 3x a Day Dose Group (N=5)
Itching two days post dose (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Itching two days post dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03843502/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03843502/ICF_001.pdf